CLINICAL TRIAL: NCT07246421
Title: Mechanisms for Glucagon Resistance as Driver of Metabolic Associated Steatotic Liver Disease and Cardiovascular Disease in Humans With Type 2 Diabetes
Brief Title: Glucagon Resistance in Patients With MASLD and T2DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MASLD_GLUCA2025; 0092321 (Other Grant/Funding Number: Steno Collaborative Grant, Novo Nordisk Foundation)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Associated Fatty Liver Disease; Type 2 Diabetes (T2DM)
Keywords: MASLD; Glucagon; Glucagon Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects with T2DM and MR spectroscopy verified NO steatosis (Active Comparator)
  Interventions: Other: Glugagon
- Subjects with T2DM and MR spectroscopy verified steatosis (Active Comparator)
  Interventions: Other: Glugagon

INTERVENTIONS:
Other: Glugagon — Infusion of low dose glucagon and high dose glucagon during simultaneous somatostatin infusion and replacement doses of insulin and growth hormone. Infusion of palmitate, VLDL-triglyceride and glucose tracers.
  [11C]palmitate PET during low and high dose glucagon.

SUMMARY:
The goal of this clinical trial is to investigate the sensitivity to glucagon in patients with type 2 diabetes mellitus (T2DM), with and without metabolic associated fatty liver disease (MASLD).

The main questions it aims to answer are:

1. Is the sensitivity to glucagon with respect to hepatic FA oxidation and suppression of VLDL-TG secretion impaired in humans with T2DM and MASLD?
2. Is glucagon resistance and MASLD reflected in an aberrated lipidomic/metabolomic profile in blood and adipose tissue?

Researchers will compare patients with T2DM with and without MASLD to see if the response to basal and high levels of glucagon differs between the groups.

Participants will attend 2 short visits and 1 full-day visit, including:

* Body scan (DXA) to check fat and bone composition
* MRI to measure liver fat.
* Blood tests.
* Ultrasound to check liver stiffness and scarring.
* Fat biopsies
* 8-hour hormone (including glucagon) and tracer infusion
* PET-CT scans

ELIGIBILITY:
Inclusion Criteria:

* BMI > 26 kg/m²
* confirmed diagnosis of Type 2 Diabetes Mellitus (T2DM) min. 6 months prior enrollment
* steatosis FF% > 5,6% on MR spectroscopy for MAFLD group

Exclusion Criteria:

* Alcohol abuse (>10 units per week for both sexes) or other substance abuse
* Smoking
* Current or previous malignant disease
* Blood donation within the last 3 months prior to the study day
* Participation in studies involving radioactive isotopes within the past 3 months
* Pregnancy
* Severely dysregulated type 2 diabetes mellitus (haemoglobin A1c ≥ 100 mmol/mol)
* C-peptide < 200 pmol/L
* Previous acute myocardial infarction (AMI)
* Clinical symptoms of heart failure
* Current or previous malignant disease
* Known ongoing systemic disease, except for dyslipidaemia and hypertension
* Regular use of medication that may affect lipid and glucose metabolism, including insulin treatment, regular use of over-the-counter medications, and hormonal contraception. Exceptions:

  1. Participants treated with statins may be included following a 2-week washout period prior to the experimental study day.
  2. Participants receiving oral glucose-lowering therapy for T2DM and antihypertensive medication may be included provided that medication is withheld on the study day only.
  3. Participants receiving weekly injectable glucagon-like peptide-1 receptor agonists (GLP-1 analogues) may be included following a 1-week washout period prior to the study day.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Hepatic FFA oxidation rate (µmol/100Ml/min) | 30 minutes at steady-state
  Measured using [11C]palmitate positron-emission tomography (PET)
Blood and adipose tissue proteomic and lipidomic profiles | 30 minutes after steady-state
  Mass spectrometry-based lipidomic/proteomic profiles of paired adipose and plasma samples.

SECONDARY OUTCOMES:
Endogen glucose production (mmol/kg/min) | 30 minutes at steady-state
  3-3H glucose tracer technique
Fatty acid turnover (µmol/min) | 30 minutesat steady-state
  Infusion af [9,10-3H] palmitate and measurement of specific activity
VLDL-triglyceride kinetics (appearance rate (µmol/min) and oxidation (µmol/min)) | 30 minutes at steady-state
  Ex vivo labeled VLDL [14C]-triolein tracer technique. Oxidation is measured by specific activity in exhaled air.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided